CLINICAL TRIAL: NCT01729520
Title: Knee Joint Pain During Strength Training After Total Knee Arthroplasty: Effect of Loading and Repetitions to Failure
Brief Title: Descriptive Study of Knee Joint Pain During Strength Training After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Bandholm, Senior Researcher, PhD, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: BA-2012-BR
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee arthroplasty; Total knee replacement; Strength training; Resistance training; Physical therapy modalities; Fatigue
MeSH Terms: conditions — Osteoarthritis, Knee; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Knee extension strength training (Experimental)
  Interventions: Other: Knee extension strength training

INTERVENTIONS:
Other: Knee extension strength training — Load experiment: Four knee extensions will be performed with the operated leg at 20, 14, and 8 RM loadings each, in a randomized order. Range of knee joint motion and time under tension for each repetition will be controlled for
  Failure experiment: One strength training set of knee extensions will be performed with the operated leg at 10 RM loading until contraction failure. Range of knee joint motion and time under tension for each repetition will be controlled for

SUMMARY:
Background:

In the early phase after a total knee arthroplasty (TKA), patients experience multi-level weakness in the operated leg, which is caused primarily by reduced central nervous system (CNS) activation failure of the muscles - especially the knee extensors. This considerable loss of muscle strength relates to reduced functional performance. Early-commenced, progressive strength training of the knee extensors of the operated leg therefore seems rational. However, the concern is that this type of early-commenced, intense physical rehabilitation exacerbates post-operative symptoms, such as knee joint pain.

The investigators have recently reported that early-commenced physical rehabilitation, including progressive strength training of the knee extensors of the operated leg seems feasible after TKA. The classic exercise-physiology literature emphasizes loading and repetitions performed to contraction failure - among others - as important variables for muscle hypertrophy and strength gains. It is currently not known how loading and repetitions performed to contraction failure during knee extensions with the operated leg, influences post-operative knee joint pain in patients with TKA.

Purpose and hypothesis:

The purpose of this study is to investigate how loading and repetitions to contraction failure influence knee joint pain during knee extensions with the operated leg early after TKA.

The hypothesis is that knee pain increases with increasing loading and fatigue.

Methods:

Fifteen patients with a unilateral TKA, operated between 1 to 2 weeks prior to the first investigation, will be included. The participants are investigated twice. During the first investigation, the absolute load (kilograms) corresponding to 10 Repetition Maximum (RM) (a load that can be lifted exactly 10 times) will be determined for unilateral (operated leg) knee extension. At the second investigation, at least 72 hours later, the patients will perform 1 set of 4 repetitions with a relative loading of 8, 14, and 20 RM each, in a randomized order, estimated from their 10 RM test at the first investigation. Time under tension (contraction velocity) and range of knee joint motion for each repetition will be controlled for. During the concentric phase of each repetition, the patients rate their knee joint pain verbally, using a numerical rating scale placed 1 meter in front of them. After a short break, the patients perform 1 set of knee extension with a relative loading of 10 RM until of contraction failure. As for the loading effect described above, they rate their knee joint pain during the concentric phase of each repetition.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral primary TKA
* Between the age of 18 to 80 years
* Understand and speak Danish
* Informed consent
* 1 to 2 weeks after TKA

Exclusion Criteria:

* Disease/Musculoskeletal disorder, which requires special rehabilitation modality
* Alcohol and drug abuse
* Lack of wish to participate or unwillingness to sign an informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Load experiment: Difference (in numerical rating scale points) between 20 RM, 14 RM, and 8 RM loadings, in knee joint pain during knee extensions. | Four repetitions at 20 RM, 14 RM, and 8 RM loadings. The strength training sets are performed at a single day, 1 to 2 weeks after surgery.
  A 0-10 numerical rating scale is used to rate knee joint pain during every repetition.
Failure experiment: Change (in numerical rating scale points) from 10% contraction failure in knee joint pain during knee extensions. | 10% to 100% contraction failure in a single strength training set performed until contraction failure. The strength training set is performed at a single day, 1 to 2 weeks after surgery.
  A 0-10 numerical rating scale is used to rate knee joint pain during every repetition.

SECONDARY OUTCOMES:
Change from baseline (pre strength training) in resting knee joint pain (numerical rating scale points). | From baseline (pre strength training) to after the strength training sets. The strength training sets are performed at a single day,1 to 2 weeks after surgery.
  A 0-10 numerical rating scale is used to rate knee joint pain at rest.
Knee joint pain (in numerical rating scale points) during activities of daily living | Before the strength training sets at a single day,1 to 2 weeks after surgery.
  Knee joint pain is rated during standing and walking, using a 0-10 numerical rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bandholm, PhD, Study Director — Clinical Research Center, Copenhagen University Hospital, Hvidovre, Copenhagen, Denmark
Locations (1):
- Clinical Research Center (136), Copenhagen University Hospital, Hvidovre, Hvidovre, Copenhagen, Denmark

REFERENCES:
- [Derived] Bandholm T, Thorborg K, Lunn TH, Kehlet H, Jakobsen TL. Knee pain during strength training shortly following fast-track total knee arthroplasty: a cross-sectional study. PLoS One. 2014 Mar 10;9(3):e91107. doi: 10.1371/journal.pone.0091107. eCollection 2014. PMID 24614574